CLINICAL TRIAL: NCT01989793
Title: A Study of Muscle Strength Maintenance in Older Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NA_00078435; P30AG021334 (NIH)
Record Dates: First submitted 2013-11-05; First posted 2013-11-21 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-06-12 (Actual); Status verified 2018-05

CONDITIONS: Sarcopenia
Keywords: sarcopenia; frailty; losartan
MeSH Terms: conditions — Sarcopenia; Frailty | interventions — Losartan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Losartan (Active Comparator): For those subjects randomized to the losartan group, they will receive losartan 25mg by mouth daily for 8 weeks, then increase to 50mg by mouth daily for another 8 weeks, then increase to 100mg by mouth daily for a final 8 weeks.
  Interventions: Drug: Losartan
- Placebo (Placebo Comparator): For those subjects randomized to placebo, they will receive a placebo to take for 24 weeks total.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Losartan — Losartan will be given in increasing doses to those in the losartan arm.
  Arms: Losartan
Drug: Placebo — Placebo will be given to those in placebo arm
  Arms: Placebo

SUMMARY:
This research study is being done to see whether losartan can prevent the decrease in strength associated with aging.

Muscle loss is associated with aging and has multiple symptoms such as weakness, slowness, and fatigue (tiredness). Older adults with muscle weakness have a higher risk of falls and disability. In addition, the loss of independence for older adults can lead to a poorer quality of life.

Recently, it was discovered that losartan, a medication commonly used to treat high blood pressure, had slowed the strength decline seen in older mice. In addition, it allowed injured mice skeletal muscle to heal faster. Therefore, we would like to see if losartan can do the same for older adults.

Losartan is approved by the Food and Drug Administration (FDA) for the treatment of high blood pressure, heart failure, and to protect the kidneys in diabetic patients. Losartan is not FDA-approved to prevent the decrease in strength associated with aging.

In this study, participants age 70 and older will be asked to take losartan or a placebo to see if losartan can help prevent loss of muscle strength. A placebo is a substance that looks like the study drug but that contains no active ingredients.

DETAILED DESCRIPTION:
The loss of independence in older adults is among the most costly and disturbing events in the life span. This loss is often influenced by multiple etiologies, including medical and neurological conditions, cognitive decline, non-supportive social/environmental settings and frailty. Frailty is a syndrome of multi-systemic, age-related decline characterized by weakness, weight loss, fatigue, low levels of activity, and slowness. Frail older adults have a higher risk for adverse outcomes including hospitalization, disability, and mortality.

Recently, Johns Hopkins University Older Americans Independence Center (JHU OAIC) investigators Burks and Cohn found that blocking angiotensin type 1 receptors with losartan, an angiotensin-receptor blocker (ARB) in older mice markedly accelerated injured skeletal muscle healing and decreased vulnerability to disuse atrophy and strength decline. These findings provide potent rationale for testing the hypothesis that losartan attenuates strength decline and other-frailty related measures in older adults.

To prepare to test this hypothesis, a phase 2 randomized, placebo controlled pilot clinical trial of losartan in pre-frail adults over age 70 is proposed that aims to assess safety and tolerability, estimate dosing range, and estimate treatment effects using inter- and intra-subject variability of potential outcome measures. Losartan is a medication that is commonly utilized in older adults for the treatment of hypertension and is generally well tolerated in that condition and in other cardiovascular conditions.

The study will take place over 24 weeks in the Clinical Research Unit (CRU) on the Hopkins Bayview Medical Campus, where 24 pre-frail subjects will be recruited from the OAIC frailty registry. Successful completion of this study will provide the safety, dosing, and outcome measure data necessary to design the pivotal study needed to determine if longer term treatment with losartan can significantly improve frailty and related skeletal muscle phenotypes.

Interventions, such as losartan, that can prevent the decline seen in frailty have the potential to improve function and help older adults maintain their independence. This is of the utmost importance in maintaining good quality-of-life for older adults.

ELIGIBILITY:
Inclusion Criteria:

* Age 70 and over
* Pre-frail as determined by frailty criteria

Exclusion Criteria:

* Under age 70
* Robust or frail by frailty criteria
* Have other indications for use of any angiotensin-receptor blockers (ARB) such as myocardial infarction in past year, history of congestive heart failure, uncontrolled hypertension
* Current use of ARBs or angiotensin-converting enzyme (ACE) inhibitors
* Prior allergic reaction to or hyperkalemia with losartan or any ARB
* Chronic renal failure with a glomerular filtration rate of < 30
* Current daily use of non-steroidal anti-inflammatory agents
* Current use of steroids
* Lower extremity disability that would prevent muscle strength testing
* Echocardiogram-diagnosed cardiac failure as evidenced by left ventricular ejection fraction less than 50%
* Cognitive impairment with a Mini-Mental State Examination < 24

Ages: 70 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Walston, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Clinical Research Unit, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Burks TN, Andres-Mateos E, Marx R, Mejias R, Van Erp C, Simmers JL, Walston JD, Ward CW, Cohn RD. Losartan restores skeletal muscle remodeling and protects against disuse atrophy in sarcopenia. Sci Transl Med. 2011 May 11;3(82):82ra37. doi: 10.1126/scitranslmed.3002227. PMID 21562229
- [Background] Abadir PM, Foster DB, Crow M, Cooke CA, Rucker JJ, Jain A, Smith BJ, Burks TN, Cohn RD, Fedarko NS, Carey RM, O'Rourke B, Walston JD. Identification and characterization of a functional mitochondrial angiotensin system. Proc Natl Acad Sci U S A. 2011 Sep 6;108(36):14849-54. doi: 10.1073/pnas.1101507108. Epub 2011 Aug 18. PMID 21852574
- [Derived] Lee JL, Zhang C, Westbrook R, Gabrawy MM, Nidadavolu L, Yang H, Marx R, Wu Y, Anders NM, Ma L, Bichara MD, Kwak MJ, Buta B, Khadeer M, Yenokyan G, Tian J, Xue QL, Siragy HM, Carey RM, de Cabo R, Ferrucci L, Moaddel R, Rudek MA, Le A, Walston JD, Abadir PM. Serum Concentrations of Losartan Metabolites Correlate With Improved Physical Function in a Pilot Study of Prefrail Older Adults. J Gerontol A Biol Sci Med Sci. 2022 Dec 29;77(12):2356-2366. doi: 10.1093/gerona/glac102. PMID 35511890
- See also: Johns Hopkins Trials listing — http://trials.johnshopkins.edu/studyData.cfm?sdUUID=C77677C9-D809-5E15-8196BB0D1BC2A829

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Losartan | Placebo
Started | 18 | 19
Completed | 10 | 15
Not Completed | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Losartan | Placebo | Total
Number analyzed (Participants) | 18 | 19 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 18 | 19 | 37
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 10 | 12 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 14 | 15 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Isokinetic Strength
Description: Isokinetic Strength was measured by knee extension exercises where bilateral knee concentric strength was measured using a Biodex System 3 dynamometer set at an angular velocity of 30deg/sec through a joint arc from 90 degrees to 30 degrees (0 degrees- full extension).
  The change in strength between baseline and week 8 (i.e., baseline minus week 8) was the outcome of the analysis. A negative number indicates that there was a decrease in isokinetic strength from week 0 to week 8.
Time Frame: Baseline to Week 8
Population: Compliant Completers: Participants who discontinued treatment during study but who continued follow-up visits and completed a final visit at 24 weeks.
Measure: Mean (Standard Deviation); unit: Newton
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 10 | 15
Newton | -4.90 (11.76) | -4.73 (8.81)
Statistical Analysis 1: Comparison: Losartan vs Placebo; Two-sample T-test of between-arm difference of change in isokinetic knee strength from baseline to week 8; Test type: Equivalence — Equivalence margin=0; p = 0.97, t-test, 2 sided

2. Primary Outcome: Change From Baseline in Isokinetic Strength
Description: Isokinetic Strength was measured by knee extension exercises where bilateral knee concentric strength was measured using a Biodex System 3 dynamometer set at an angular velocity of 30deg/sec through a joint arc from 90 degrees to 30 degrees (0 degrees- full extension).
  The change in strength between baseline and week 16 (i.e., baseline minus week 16) was the outcome of the analysis. A negative number indicates decrease in strength from week 0 to week 16.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Newton
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 10 | 15
Newton | -7.40 (9.56) | -4.27 (11.54)
Statistical Analysis 1: Comparison: Losartan vs Placebo; Two-sample T-test of between-arm difference of change in isokinetic knee strength from baseline to week 16; Test type: Equivalence — Equivalence margin=0; p = 0.48, t-test, 2 sided

3. Primary Outcome: Change From Baseline in Isokinetic Strength
Description: Isokinetic Strength was measured by knee extension exercises where bilateral knee concentric strength was measured using a Biodex System 3 dynamometer set at an angular velocity of 30deg/sec through a joint arc from 90 degrees to 30 degrees (0 degrees- full extension).
  The change in strength between baseline and week 24 (i.e., baseline minus week 24) was the outcome of the analysis. A negative number indicates a decrease in strength from week 0 to week 24.
Time Frame: Baseline to Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Newton
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 10 | 15
Newton | -9.20 (8.94) | -7.00 (10.24)
Statistical Analysis 1: Comparison: Losartan vs Placebo; Two-sample T-test of between-arm difference of change in isokinetic knee strength from baseline to week 24; Test type: Equivalence — Equivalence margin = 0; p = 0.59, t-test, 2 sided

4. Primary Outcome: Fatiguability
Description: Fatiguability was tested using bilateral knee extension with an external load equal to 40% of the maximal voluntary contraction force.
  Fatiguability was defined as the ratio (expressed as a percentage) of the total work in the last 3 of the 10 repetitions to the total work in the first 3 of the 10 repetitions, where the total work for n repetitions is defined as the sum of peak torque (FT-LBS) over n repetitions (i.e., last three reps/first three reps). The maximum of the two sides was used in the analysis.
Time Frame: Week 8
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of work
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 10 | 15
percentage of work | 14.29 (9.65) | 7.87 (15.31)
Statistical Analysis 1: Comparison: Losartan vs Placebo; Two-sample T-test of between-arm difference in fatiguability at week 8; Test type: Equivalence — Equivalence margin=0; p = 0.212, t-test, 2 sided; assuming unequal variance between arms

5. Primary Outcome: Fatiguability
Description: Fatiguability was tested using bilateral knee extension with an external load equal to 40% of the maximal voluntary contraction force.
  Fatiguability was defined as the ratio (expressed as a percentage) of the total work in the last 3 of the 10 repetitions to that of the first 3 of the 10 repetitions, where the total work for n repetitions is defined as the sum of peak torque (FT-LBS) over n repetitions (i.e., last three reps/first three reps). The maximum of the two sides was used in the analysis.
Time Frame: Week 16
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of work
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 10 | 15
percentage of work | 16.51 (18.92) | 8.77 (12.15)
Statistical Analysis 1: Comparison: Losartan vs Placebo; Two-sample T-test of between-arm difference in fatiguability at week 16; Test type: Equivalence — Equivalence margin=0; p = 0.271, t-test, 2 sided; assuming unequal variance between arms

6. Primary Outcome: Fatiguability
Description: as for outcome 5
Time Frame: Week 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of work
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 10 | 15
percentage of work | 17.07 (15.34) | 9.05 (14.15)
Statistical Analysis 1: Comparison: Losartan vs Placebo; Two-sample T-test of between-arm difference in fatiguability at week 24; Test type: Equivalence — Equivalence margin=0; p = 0.203, t-test, 2 sided; assuming unequal variance between arms

7. Secondary Outcome: Number of Participants Experiencing Any Amount of Decrease in Frailty
Description: Number of participants experiencing any amount of decrease in frailty score from baseline to Week 8 (i.e., improvement in frailty status)
Time Frame: from baseline to 8 weeks
Population: Compliant completers: participants who continued treatment during the entire 24 week study. and completed the final visit at 24 weeks. 10 out of the 18 participant who were given losartan completed the study and 15 out of 19 who received the placebo participant completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 10 | 15
Participants | 3 | 6
Statistical Analysis 1: Comparison: Losartan vs Placebo; Fisher's exact test of percentage of participants with improvement in frailty score from baseline between treatment and placebo arms; Test type: Equivalence — Equivalence margin = 0; p = 0.82, Fisher Exact

8. Secondary Outcome: Number of Participants Experiencing Any Amount of Decrease in Frailty
Description: Number of participants experiencing any amount of decrease in frailty score from baseline to Week 16 (i.e., improvement in frailty status)
Time Frame: from baseline to 16 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 10 | 15
Participants | 3 | 5
Statistical Analysis 1: Comparison: Losartan vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Equivalence — Equivalence margin = 0; p = 0.73, Fisher Exact

9. Secondary Outcome: Number of Participants Experiencing Any Amount of Decrease in Frailty
Description: Number of participants experiencing any amount of decrease in frailty score from baseline to Week 24 (i.e., improvement in frailty status)
Time Frame: from baseline to 24 weeks
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Losartan | Placebo
Number analyzed (Participants) | 10 | 15
Participants | 3 | 5
Statistical Analysis 1: Comparison: Losartan vs Placebo; [analysis description as in outcome 7, analysis 1]; Test type: Equivalence — Equivalence margin = 0; p = 0.73, Fisher Exact

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Losartan | Placebo
All-Cause Mortality (participants affected / at risk) | 1/18 | 0/19
Serious Adverse Events (participants affected / at risk) | 1/18 | 0/19
Other Adverse Events (participants affected / at risk) | 4/18 | 0/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=18) | Placebo (N=19)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Losartan (N=18) | Placebo (N=19)
Fatigue (General disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Creatinine (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes